CLINICAL TRIAL: NCT00069901
Title: CT-2103/Carboplatin for Patients With Newly Diagnosed Stage III or IV Ovarian or Primary Peritoneal Cancer: A Phase 2 Study
Brief Title: Phase II CT-2103/Carboplatin in Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGT201
Record Dates: First submitted 2003-10-02; First posted 2003-10-06 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Ovarian Neoplasm
Keywords: ovarian cancer; paclitaxel; carboplatin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — paclitaxel poliglumex; Carboplatin

INTERVENTIONS:
Drug: CT-2103 (poly(L)glutamate-paclitaxel)
Drug: carboplatin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of CT-2103 (poly(L)glutamate-paclitaxel) in combination with carboplatin for the treatment of patients with Stage III or IV ovarian or primary peritoneal cancer.

DETAILED DESCRIPTION:
CT-2103 is a pharmaceutical that links paclitaxel, the active ingredient in Taxol(R), to a biodegradable polyglutamate polymer. The objective of this trial is to evaluate the toxicity, estimate the response rate, progression-free survival and overall survival in patients with newly diagnosed stage III or IV ovarian or primary peritoneal carcinoma treated with CT-2103 in combination with carboplatin.

ELIGIBILITY:
Inclusion criteria:

* Histologically-confirmed stage III or IV ovarian carcinoma or primary peritoneal cancer patients who have had appropriate debulking surgery for ovarian or peritoneal carcinoma.
* Patients must be recovered from initial surgery and must enter this study no later than 12 weeks after such surgery.
* ECOG performance score of 0, 1, or 2.
* absolute neutrophil count (ANC) at least 1,500/µL.
* platelet at least 100,000/µL.
* hemoglobin at least 10 g/dL.
* creatinine no greater than 1.5 times the upper limit of normal (ULN).
* bilirubin no greater than 1.5 x ULN (if liver metastases are not present, SGOT and SGPT no greater than 2.5 x ULN, if liver metastases are present, SGOT and SGPT may be no greater than 5 x ULN.
* Alkaline phosphatase no greater than 2.5 x ULN.

Exclusion:

* Current diagnosis of epithelial ovarian tumor of low malignant potential (borderline carcinomas)
* Germ cell tumors, sex cord-stromal tumors, carcinosarcomas, mixed mullerian tumors or carcinosarcomas, metastatic carcinomas from sites other than the ovary, and low malignant potential tumors including so called micropapillary serous carcinomas.
* Synchronous primary endometrial cancer or history of primary endometrial cancer.
* Evidence of any other invasive malignancies present within the 3 years before this study, with the exception of non-melanoma skin cancer and other specific malignancies as noted above.
* Any prior treatment, other than initial debulking surgery, for the cancer being treated in this study.
* Patients may have received prior adjuvant chemotherapy for localized breast cancer, if the therapy was completed at least 3 years before registration in this study and if the patient remains free of recurrent or metastatic disease.
* Prior radiotherapy to any portion of the abdominal cavity or pelvis.
* Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, if it was completed at least 3 years before registration in this study and if the patient remains free of recurrent or metastatic disease.
* Administration of other investigational drugs within 26 weeks before the first treatment in this study. Toxic manifestations of previous treatments (except alopecia) must have been stable for 4 weeks.
* Presence of active hepatitis, either acute or chronic.
* Presence of active infection requiring antibiotic or antiviral therapy.
* Pregnant women or nursing mothers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2003-02; Primary Completion 2005-11 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Stromatt, M.D., Study Director — CTI BioPharma
Locations (17):
- United States (17):
  - California Cancer Care, Greenbrae, California
  - Gynecology Oncology Associates, Greenbrae, California
  - Stockton Hematology Oncology Medical, Stockton, California
  - Raben and Fldman Research Associates, South Miami, Florida
  - University of Louisville, Louisville, Kentucky
  - Resource Center for Gynecology/ Oncology, Kansas City, Missouri
  - Upstate New York Cancer Research and Education Foundation, Rochester, New York
  - Gynecology, Oncology, and Pelvic Surgery Associates, Inc., Columbus, Ohio
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - South Carolina Oncology Assoicates, Columbia, South Carolina
  - Chattanooga GYN-Oncology, Chattanooga, Tennessee
  - Baptist Regional Cancer Center, Knoxville, Tennessee
  - Arlington Fairfax Hematology Oncology, Arlington, Virginia
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Aurora Health Care, Inc., Milwaukee, Wisconsin